CLINICAL TRIAL: NCT00364156
Title: Comparison of Standard Versus Extended Nicotine Patch Therapy for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 801851; P50CA084718 (NIH)
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Results first posted 2010-11-02 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: TOBACCO USE CESSATION
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended Patch Treatment (Experimental): Participants in this treatment arm receive 24 weeks of 21mg nicotine patch in addition to 8 smoking cessation counseling sessions.
  Interventions: Drug: 24-weeks of nicotine patch
- Standard Patch Treatment (Active Comparator): Participants receive 8 weeks of 21mg nicotine patch followed by 16 weeks of placebo patch.
  Interventions: Drug: Standard Patch Treatment

INTERVENTIONS:
Drug: Standard Patch Treatment — 8-weeks of nicotine patch + 16-weeks of placebo
  Arms: Standard Patch Treatment
Drug: 24-weeks of nicotine patch — 24-weeks of 21mg nicotine patch
  Arms: Extended Patch Treatment

SUMMARY:
This randomized double-blind, placebo-controlled will determine the relative efficacy of standard versus extended transdermal nicotine (TN) therapy for smoking cessation. After completing the eligibility screening, 600 treatment-seeking smokers will be randomized to receive either standard treatment (ST) with TN (21mg x 8 weeks, placebo x 16 weeks) or extended treatment (ET) with TN (21mg x 24 weeks). All participants will receive behavioral counseling. The primary outcome will be biochemically verified abstinence from smoking at the end of treatment (week 24). Secondary outcomes include abstinence at week 28 (4 weeks after treatment is discontinued), and time to failure. We hypothesize that ET will produce significantly higher quit rates than ST; however, the benefit of ET will last only so long as treatment is continued. Support for this hypothesis would indicate that maintenance therapy with TN should be considered.

DETAILED DESCRIPTION:
Please see brief summary.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of descent between the ages of 18-65 who smokes at least 10 cigarettes/day and are seeking smoking cessation treatment.
2. Based on the medical history, physical and laboratory examination, premenopausal female subjects must consent to practice an effective form of contraception during study.
3. Following orientation by the research staff, subjects must sign written informed consent for all study procedures.

Exclusion Criteria:

1. Women who are pregnant, planning a pregnancy, or lactating.
2. Current medical problems for which TN is contraindicated including allergy to nicotine, uncontrolled hypertension, unstable angina, serious arrhythmia, heart attack or stroke within the past 6 months, liver and/or kidney failure in the last 6-months and current diabetes.
3. Current treatment of cancer or diagnosed with cancer in the past 6 months
4. Current DSM IV substance use disorders (dependence involving alcohol, cocaine, marijuana or stimulants, benzodiazepines).
5. Current use of TN or other forms of NRT.
6. Concomitant medications (e.g., monoamine oxidase inhibitors or benzodiazepines within past 14 days, antipsychotics, endogenous steroids, and antidepressants (including wellbutrin or bupropion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2004-06; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Tobacco Use Research Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Patterson F, Kerrin K, Wileyto EP, Lerman C. Increase in anger symptoms after smoking cessation predicts relapse. Drug Alcohol Depend. 2008 May 1;95(1-2):173-6. doi: 10.1016/j.drugalcdep.2008.01.013. Epub 2008 Mar 6. PMID 18328642
- [Result] Schnoll RA, Patterson F, Wileyto EP, Heitjan DF, Shields AE, Asch DA, Lerman C. Effectiveness of extended-duration transdermal nicotine therapy: a randomized trial. Ann Intern Med. 2010 Feb 2;152(3):144-51. doi: 10.7326/0003-4819-152-3-201002020-00005. PMID 20124230
- [Result] Schnoll RA, Patterson F, Wileyto EP, Tyndale RF, Benowitz N, Lerman C. Nicotine metabolic rate predicts successful smoking cessation with transdermal nicotine: a validation study. Pharmacol Biochem Behav. 2009 Mar;92(1):6-11. doi: 10.1016/j.pbb.2008.10.016. Epub 2008 Oct 31. PMID 19000709
- [Result] Lerman C, Jepson C, Wileyto EP, Patterson F, Schnoll R, Mroziewicz M, Benowitz N, Tyndale RF. Genetic variation in nicotine metabolism predicts the efficacy of extended-duration transdermal nicotine therapy. Clin Pharmacol Ther. 2010 May;87(5):553-7. doi: 10.1038/clpt.2010.3. Epub 2010 Mar 24. PMID 20336063
- [Result] Ray R, Mitra N, Baldwin D, Guo M, Patterson F, Heitjan DF, Jepson C, Wileyto EP, Wei J, Payne T, Ma JZ, Li MD, Lerman C. Convergent evidence that choline acetyltransferase gene variation is associated with prospective smoking cessation and nicotine dependence. Neuropsychopharmacology. 2010 May;35(6):1374-82. doi: 10.1038/npp.2010.7. Epub 2010 Feb 10. PMID 20147892
- [Derived] Ashare RL, Wileyto EP, Perkins KA, Schnoll RA. The first 7 days of a quit attempt predicts relapse: validation of a measure for screening medications for nicotine dependence. J Addict Med. 2013 Jul-Aug;7(4):249-54. doi: 10.1097/ADM.0b013e31829363e1. PMID 23669629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using mass media advertising from the the Greater Philadelphia area from June 2004 to April 2008.
Pre-assignment Details: Once participants were enrolled and were eligible at the medical screening visit they were randomized to receiving either 8 weeks of 21 mg nicotine patch or 6 months of 21 mg nicotine patch treatment
Groups:
- Extended Patch Treatment: Participants in this treatment arm receive 24 weeks of 21 mg nicotine patch in addition to 8 smoking cessation counseling sessions.
- Standard Patch Treatment: Participants receive 8 weeks of 21 mg nicotine patch followed by 16 weeks of placebo patch.
Period: Overall Study
Arm/Group | Extended Patch Treatment | Standard Patch Treatment
Started | 282 | 286
Completed | 203 | 205
Not Completed | 79 | 81
Not completed — Withdrawal by Subject | 73 | 80
Not completed — Protocol Violation | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Patch Treatment | Standard Patch Treatment | Total
Number analyzed (Participants) | 282 | 286 | 568
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 281 | 286 | 567
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (10.2) | 44.9 (10.4) | 44.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 129 | 254
  Male | 157 | 157 | 314
Region of Enrollment [Number; unit: participants]
  United States | 282 | 286 | 568

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Verified 7-day Point Prevalence Abstinence
Description: To evaluate the efficacy of standard (8-week) vs. extended (24-week) transdermal nicotine therapy.
Time Frame: End of Treatment (week 24)
Population: Intention to Treat analysis (ITT)
Measure: Number; unit: Participants
Arm/Group | Extended Patch Treatment | Standard Patch Treatment
Number analyzed (Participants) | 282 | 286
Participants | 89 | 58

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Extended Patch Treatment | Standard Patch Treatment
Serious Adverse Events (participants affected / at risk) | 0/282 | 1/286
Other Adverse Events (participants affected / at risk) | 4/282 | 0/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Patch Treatment (N=282) | Standard Patch Treatment (N=286)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — 10/4/2007: Participant disclosed that she had recently had a stroke shortly after her last visit to the center. She sought medical attention immediately and was advised by her physician to discontinue use of the nicotine patch.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Patch Treatment (N=282) | Standard Patch Treatment (N=286)
Agressive Thoughts (Psychiatric disorders) | 1 (1) | 0 (0) — 10/23/2007-During Session 2 of the study participant reported feeling distraught & aggressive thoughts towards family members due to certain personal circumstances. Case discussed & participant provided with mental health helpline & other resources.
Seizure during Blood Draw (Nervous system disorders) | 1 (1) | 0 (0) — 4/17/2006: Participant had a 30-40 sec seizure after their blood draw. Participant recovered on their own from the seizure. Participant was monitored & their vitals were normal. Participants successfully completed rest of the session feeling normal
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) — 2 Participants had high BP readings >200/110 during participating in the study. Both participants were encouraged to received medical help for uncontrolled hypertension, and discontinue nicotine patch treatment and only receive counseling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No